CLINICAL TRIAL: NCT00087516
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of MK0431 Monotherapy in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: Monotherapy Study in Patients With Type 2 Diabetes Mellitus (0431-021)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-021; Formally-C0604MT2D; MK0431-021; 2006_413
Record Dates: First submitted 2004-07-09; First posted 2004-07-13 (Estimated); Results first posted 2010-06-08 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Sitagliptin 100 mg/100 mg (Active Comparator): Phase A and B: Oral tablets of sitagliptin 100 mg Once a Day (q.d )
  Interventions: Drug: Sitagliptin (MK0431); Drug: Metformin - Rescue
- Sitagliptin 200 mg/200 mg (Active Comparator): Phase A and B: Oral tablets of sitagliptin 200 mg q.d
  Interventions: Drug: Sitagliptin; Drug: Metformin - Rescue
- Placebo/Sitagliptin 100 mg (Placebo Comparator): Phase A: Oral tablets of placebo matching sitagliptin 100 mg q.d. Phase B: Oral tablets of sitagliptin 100 mg q.d.
  Interventions: Drug: Placebo; Drug: Metformin - Rescue
- Placebo/Sitagliptin 200 mg (Placebo Comparator): Phase A: Oral tablets of placebo matching sitagliptin 200 mg q.d. Phase B: Oral tablets of sitagliptin 200 mg q.d.
  Interventions: Drug: Placebo; Drug: Metformin - Rescue

INTERVENTIONS:
Drug: Sitagliptin (MK0431) — Phase A: Sitagliptin 100 mg once a day for 24 weeks. Phase B: Sitagliptin 100 mg once a day for 80 weeks.
  Other Names: MK0431; Januvia
  Arms: Sitagliptin 100 mg/100 mg
Drug: Sitagliptin — Phase A: Sitagliptin 200 mg once a day for 24 weeks. Phase B: Sitagliptin 200 mg once a day for 80 weeks.
  Other Names: MK0431; Januvia
  Arms: Sitagliptin 200 mg/200 mg
Drug: Placebo — Phase A: Placebo matching Sitagliptin 100 mg once a day for 24 weeks. Phase B: Sitagliptin 100 mg once a day for 80 weeks.
  Arms: Placebo/Sitagliptin 100 mg
Drug: Placebo — Phase A: Placebo matching Sitagliptin 200 mg once a day for 24 weeks. Phase B: Sitagliptin 200 mg once a day for 80 weeks.
  Arms: Placebo/Sitagliptin 200 mg
Drug: Metformin - Rescue — Phase A: Patients not meeting specific glycemic goals will receive open-label metformin as 500 mg, 850 mg, and 1000 mg oral tablets titrated at the discretion of the investigator. Phase B: These patients will not initiate Phase B double-blind medication.
  Other Names: Metformin; Glucophage; Glucophage XR; Glumetza; Fortamet; Riomet

SUMMARY:
The purpose of this clinical study is to determine the safety and efficacy of an investigational drug in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* Patient is not pregnant or breastfeeding
* Male or female patient unlikely to conceive
* Patient not on an antihyperglycemic drug

Exclusion Criteria:

* Patient has history of type 1 diabetes mellitus
* Patient has history of ketoacidosis
* Patient requires insulin within 8 weeks prior to start of study
* Patient on weight loss program and is not in maintenance phase
* Patient taking weight loss medication within 8 weeks prior to start of study
* Patient on or likely to require = 14 days or repeated courses of corticosteroids
* Patient taking immunosuppressive/immunomodulating medication
* Patient taking digoxin or other cardiac medication
* Patient has undergone surgical general anesthesia within 30 days prior to start of study
* Patient taking investigational drug within 8 weeks prior to start of study
* Patient is diagnosed with liver disease
* Patient has chronic myopathy, progressive neurological/neuromuscular disorder
* Patient has with severe cardiac conditions within the last 6 months
* Patient is Human immunodeficiency virus (HIV) positive
* Patient has hematological disorder
* Patient has history of malignancy
* Patient has history of alcohol or drug abuse within the past 3 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2004-06; Primary Completion 2005-07 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Aschner P, Kipnes MS, Lunceford JK, Sanchez M, Mickel C, Williams-Herman DE; Sitagliptin Study 021 Group. Effect of the dipeptidyl peptidase-4 inhibitor sitagliptin as monotherapy on glycemic control in patients with type 2 diabetes. Diabetes Care. 2006 Dec;29(12):2632-7. doi: 10.2337/dc06-0703. PMID 17130196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 08-Jul-2004; Last Patient Last Visit: 07-Feb-2007; One hundred eleven medical clinics worldwide (56 in the United States and Puerto Rico, 16 in 6 countries in Europe and 39 in 11 countries in the rest of the world).
Pre-assignment Details: Patients 18-75 years not on an antihyperglycemic agent (AHA) or on oral single AHA or low-dose combination therapy were eligible to participate. Following a screening diet/exercise period of variable duration, patients with hemoglobin A1c (A1C) 7-10% were eligible to enter a 2-week placebo run-in/wash-off period prior to randomization.
Groups:
- Sitagliptin 100 mg/100 mg: The Sitagliptin 100 mg/100 mg group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 100 mg q.d. (once daily) for up to 104 weeks (including the 24-week Phase A study period and 80-week Phase B study period).
- Sitagliptin 200 mg/200 mg: The Sitagliptin 200 mg/200 mg group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 200 mg q.d. for up to 104 weeks (including the 24-week Phase A study period and 80-week Phase B study period).
- Placebo/Sitagliptin 100 mg: The Placebo/Sitagliptin 100 mg group includes data from patients randomized to receive treatment with oral tablets of sitagliptin-matching placebo tablets once daily during the 24-week Phase A study period followed by oral tablets of sitagliptin 100 mg q.d. during the 80-week Phase B study period.
- Placebo/Sitagliptin 200 mg: The Placebo/Sitagliptin 200 mg group includes data from patients randomized to receive treatment with oral tablets of sitagliptin-matching placebo tablets once daily during the 24-week Phase A study period followed by oral tablets of sitagliptin 200 mg q.d. during the 80-week Phase B study period.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg/100 mg | Sitagliptin 200 mg/200 mg | Placebo/Sitagliptin 100 mg | Placebo/Sitagliptin 200 mg
Started | 238 | 250 | 130 | 123
Completed | 77 | 81 | 33 | 38
Not Completed | 161 | 169 | 97 | 85
Not completed — Adverse Event | 10 | 10 | 3 | 6
Not completed — Lack of Efficacy | 82 | 80 | 39 | 29
Not completed — Lost to Follow-up | 8 | 6 | 5 | 5
Not completed — Protocol Violation | 4 | 8 | 3 | 6
Not completed — Withdrawal by Subject | 16 | 27 | 11 | 12
Not completed — Site terminated | 0 | 2 | 1 | 0
Not completed — Protocol specified discontinuation | 35 | 33 | 33 | 26
Not completed — Patient moved | 3 | 2 | 1 | 0
Not completed — Patient was non-compliant | 3 | 1 | 0 | 0
Not completed — Recommendation of Primary Care Physician | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin 100 mg: The Sitagliptin 100 mg/100 mg group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 100 mg q.d. (once daily) for up to 104 weeks (including the 24-week Phase A study period and 80-week Phase B study period).
- Sitagliptin 200 mg: The Sitagliptin 200 mg/200 mg group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 200 mg q.d. for up to 104 weeks (including the 24-week Phase A study period and 80-week Phase B study period).
- Placebo: The Placebo group includes data from patients randomized to receive treatment with oral tablets of sitagliptin-matching placebo tablets once daily during the 24-week Phase A study period followed by oral tablets of sitagliptin 100 or 200 mg q.d. during the 80-week Phase B study period.
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo | Total
Number analyzed (Participants) | 238 | 250 | 253 | 741
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (9.5) | 54.9 (10.1) | 54.3 (10.1) | 54.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 133 | 123 | 358
  Male | 136 | 117 | 130 | 383
Race/Ethnicity, Customized [Number; unit: participants]
  White | 122 | 132 | 127 | 381
  Black | 10 | 12 | 16 | 38
  Hispanic | 58 | 53 | 64 | 175
  Asian | 32 | 37 | 34 | 103
  Other | 16 | 16 | 12 | 44
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 170.7 (43.0) | 174.2 (46.2) | 176.1 (41.8) | 173.7 (43.7)
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] | 8.0 (0.9) | 8.1 (0.9) | 8.0 (0.8) | 8.0 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: A1C is measured as a percent. Thus, this change from baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent.
Time Frame: Weeks 0-24
Population: The all-patients-treated population included all patients with at least one dose of double-blind study therapy, and with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. Missing data were handled using the last observation carrying forward method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo
Number analyzed (Participants) | 229 | 238 | 244
Percent | -0.61 [-0.74 to -0.49] | -0.76 [-0.88 to -0.64] | 0.18 [0.06 to 0.30]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, presence/absence of prior diabetes pharmacotherapy, baseline A1C; Mean Difference (Net) = -0.79, 95% CI [-0.96 to -0.62], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Sitagliptin 200 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, presence/absence of prior diabetes pharmacotherapy, baseline A1C; Mean Difference (Net) = -0.94, 95% CI [-1.11 to -0.77], Standard Error of Mean 0.09

2. Secondary Outcome: Change From Baseline in FPG at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 FPG minus Week 0 FPG.
Time Frame: Weeks 0-24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo
Number analyzed (Participants) | 234 | 244 | 247
mg/dL | -12.4 [-17.4 to -7.4] | -16.6 [-21.5 to -11.7] | 4.7 [-0.2 to 9.6]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, presence/absence of prior diabetes pharmacotherapy, baseline FPG; Mean Difference (Net) = -17.1, 95% CI [-24.1 to -10.1], Standard Error of Mean 3.6
Statistical Analysis 2: Comparison: Sitagliptin 200 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, presence/absence of prior diabetes pharmacotherapy, baseline FPG; Mean Difference (Net) = -21.3, 95% CI [-28.2 to -14.4], Standard Error of Mean 3.5

3. Secondary Outcome: Change From Baseline in 2-hour Post-meal Glucose (2-hr PMG) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 2-hr PMG minus Week 0 2-hr PMG.
Time Frame: Weeks 0-24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo
Number analyzed (Participants) | 201 | 205 | 204
mg/dL | -48.9 [-57.9 to -40.0] | -56.3 [-65.2 to -47.5] | -2.2 [-11.1 to 6.7]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, presence/absence of prior diabetes pharmacotherapy, baseline 2-hr PMG; Mean Difference (Net) = -46.7, 95% CI [-59.4 to -34.1], Standard Error of Mean 6.5
Statistical Analysis 2: Comparison: Sitagliptin 200 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, presence/absence of prior diabetes pharmacotherapy, baseline 2-hr PMG; Mean Difference (Net) = -54.1, 95% CI [-66.7 to -41.6], Standard Error of Mean 6.4

4. Secondary Outcome: Change From Baseline in A1C at Week 104
Description: A1C is measured as a percent. Thus, this change from baseline reflects the Week 104 A1C percent minus the Week 0 A1C percent.
Time Frame: Weeks 0-104
Population: The all-patients-treated population for Week 104 included all patients with at least one dose of double-blind study therapy after Week 24, and with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. Missing data were handled using the last observation carrying forward method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Placebo/ Sitagliptin 100 mg: The Placebo/Sitagliptin 100 mg group includes data from patients randomized to receive treatment with oral tablets of sitagliptin-matching placebo tablets once daily during the 24-week Phase A study period followed by oral tablets of sitagliptin 100 mg q.d. during the 80-week Phase B study period.
Arm/Group | Sitagliptin 100 mg/100 mg | Sitagliptin 200 mg/200 mg | Placebo/ Sitagliptin 100 mg | Placebo/Sitagliptin 200 mg
Number analyzed (Participants) | 188 | 195 | 81 | 83
Percent | -0.27 [-0.41 to -0.13] | -0.40 [-0.53 to -0.26] | -0.32 [-0.53 to -0.11] | -0.34 [-0.55 to -0.13]

5. Secondary Outcome: Change From Baseline in FPG at Week 104
Description: Change from baseline at Week 104 is defined as Week 104 FPG minus Week 0 FPG.
Time Frame: Weeks 0-104
Population: The all-patients-treated population for Week 104, included all patients with at least one dose of double-blind study therapy after Week 24, and with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. Missing data were handled using the last observation carrying forward method.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg/100 mg | Sitagliptin 200 mg/200 mg | Placebo/Sitagliptin 100 mg | Placebo/Sitagliptin 200 mg
Number analyzed (Participants) | 190 | 194 | 81 | 83
mg/dL | -1.8 [-7.3 to 3.7] | -5.7 [-11.1 to -0.2] | -4.1 [-12.5 to 4.3] | -4.1 [-12.4 to 4.2]

6. Secondary Outcome: Change From Baseline in 2-hr PMG at Week 104
Description: Change from baseline at Week 104 is defined as Week 104 2-hr PMG minus Week 0 2-hr PMG.
Time Frame: Weeks 0-104
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg/100 mg | Sitagliptin 200 mg/200 mg | Placebo/Sitagliptin 100 mg | Placebo/Sitagliptin 200 mg
Number analyzed (Participants) | 165 | 168 | 68 | 63
mg/dL | -30.5 [-40.1 to -21.0] | -41.5 [-51.0 to -32.1] | -38.3 [-53.2 to -23.4] | -35.5 [-50.9 to -20.1]

ADVERSE EVENTS:
Time Frame: Weeks 0-104
Arm/Group | Sitagliptin 100 mg/100 mg | Sitagliptin 200 mg/200 mg | Placebo/Sitagliptin 100 mg | Placebo/Sitagliptin 200 mg
Serious Adverse Events (participants affected / at risk) | 24/238 | 25/250 | 10/130 | 13/123
Other Adverse Events (participants affected / at risk) | 127/238 | 137/250 | 70/130 | 65/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg/100 mg (N=238) | Sitagliptin 200 mg/200 mg (N=250) | Placebo/Sitagliptin 100 mg (N=130) | Placebo/Sitagliptin 200 mg (N=123)
Angina Pectoris (Cardiac disorders) | 2 | 1 | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 3
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Borderline Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Gallbladder Necrosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 1 | 2
Abscess Of Salivary Gland (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis Acute (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia Legionella (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Urethritis (Infections and infestations) | 1 | 0 | 0 | 0
Anaesthetic Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foreign Body Trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lung Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radial Nerve Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0 | 0
Lipase Increased (Investigations) | 1 | 0 | 0 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adrenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Benign Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung Adenocarcinoma Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Lacunar Infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0 | 0
Suicidal Behavior (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vaginal Cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg/100 mg (N=238) | Sitagliptin 200 mg/200 mg (N=250) | Placebo/Sitagliptin 100 mg (N=130) | Placebo/Sitagliptin 200 mg (N=123)
Constipation (Gastrointestinal disorders) | 14 | 11 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 17 | 17 | 3 | 7
Nausea (Gastrointestinal disorders) | 7 | 13 | 3 | 2
Influenza (Infections and infestations) | 13 | 22 | 8 | 11
Nasopharyngitis (Infections and infestations) | 21 | 19 | 12 | 11
Sinusitis (Infections and infestations) | 7 | 16 | 5 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 36 | 41 | 17 | 14
Urinary Tract Infection (Infections and infestations) | 14 | 18 | 5 | 5
Blood Glucose Increased (Investigations) | 15 | 14 | 10 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 14 | 6 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 16 | 11 | 6
Dizziness (Nervous system disorders) | 25 | 31 | 15 | 10
Headache (Nervous system disorders) | 19 | 17 | 8 | 8
Hypertension (Vascular disorders) | 10 | 15 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.